CLINICAL TRIAL: NCT01804192
Title: Is Acupoints Sensation Necessary for Acu-TENS to Elicit Physiological Changes in Healthy Subjects?
Acronym: Acu-TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Yu Tai Wai David, Principle investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20080514001
Record Dates: First submitted 2013-02-11; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Autonomic Nervous System Disorder
Keywords: Acu-TENS; MAP; HR; HRV
MeSH Terms: conditions — Primary Dysautonomias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acu-TENS to LI4 and LI11 (Experimental): Acu-TENS Group (Experimental Group), subjects received TENS over right L14 and LI11.
  Systolic and diastolic blood pressures will be taken on the left arm by a digital blood pressure monitor. The mean arterial pressure (MAP) will be recorded from the machine. Three ECG electrodes will be applied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device. The heart rate (HR) will be measured. The ECG signals will be transferred to the PowerLab 16/30 for data acquisition and analysis of the HRV.
  Interventions: Other: Acu-TENS
- Control group (Active Comparator): Control Acu-TENS Group (Control Group), subjects received TENS over tips of bilateral knee caps.
  Systolic and diastolic blood pressures will be taken on the left arm by a digital blood pressure monitor. The mean arterial pressure (MAP) will be recorded from the machine. Three ECG electrodes will be applied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device. The heart rate (HR) will be measured. The ECG signals will be transferred to the PowerLab 16/30 for data acquisition and analysis of the HRV.
  Interventions: Other: Acu-TENS
- Placebo group (Placebo Comparator): Placebo Acu-TENS Group (Placebo Group), subjects received the same protocol as the Acu-TENS group and TENS was applied over right LI4 and LI11 that covered with non-conducting plastics (with the same dimension as the TENS electrodes) Systolic and diastolic blood pressures will be taken on the left arm by a digital blood pressure monitor. The mean arterial pressure (MAP) will be recorded from the machine. Three ECG electrodes will be applied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device. The heart rate (HR) will be measured. The ECG signals will be transferred to the PowerLab 16/30 for data acquisition and analysis of the HRV.
  Interventions: Other: Acu-TENS

INTERVENTIONS:
Other: Acu-TENS — Systolic and diastolic blood pressures will be taken on the left arm by a digital blood pressure monitor (Mindray PM-8000 Express Patient Monitor, Bio-Medical Electricity, Hamburg, Germany). The mean arterial pressure (MAP) will be recorded from the machine. Three ECG electrodes will be applied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device (Mindray PM-8000 Express Patient Monitor, Bio-Medical Electricity, Hamburg, Germany). The heart rate (HR) will be measured. The ECG signals will be transferred to the PowerLab 16/30 (ADInstruments Pty Ltd. NSW, Australia) for data acquisition and analysis of the HRV.
  Other Names: A dual channel portable TENS unit

SUMMARY:
Traditional Chinese Medicine (TCM) practitioners believe that health can be maintained if the body has a balanced ying-yang or the qi flows in correct strength and quality along the meridians.Stimulation of the acupoints such as by acupuncture can awaken and modulate qi in the channels and is able to regulate and restore yin-yang balance.However, there are some drawbacks associated with acupuncture which may limit its applications. These include transmission of infectious disease, pneumothorax and other problems associated with organ punctures, cardiac tamponade, and broken needles with remnants migrating to other locations.Studies have shown that when TENS is applied over acupoints (Acu-TENS), it is effective in reducing dyspnoea in patients with chronic obstructive pulmonary disease,facilitate early haemodynamic recovery after open-heart surgery,relieve labor pain,increase in blood β-endorphin level,reduce blood pressure changes in normal healthy subjects and decrease airway resistance.Despite these promising results, how Acu-TENS works still remain unclear.This study aimed to investigate the effects of Acu-TENS over Hegu (LI4) and Quichi (LI4) on the autonomic nervous system activities and to investigate whether the subject could experience distinct sensation as deqi.

DETAILED DESCRIPTION:
Eligibility criteria: Normal healthy subjects who were naïve to Acu-TENS and able to read Chinese.

Outcome Measures: Heart rate, Mean arterial blood pressure, Heart rate variability

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy subjects who were naïve to Acu-TENS and able to read Chinese were recruited for study

Exclusion Criteria:

* history of cardiopulmonary, neurological and psychologic disorders or they required taking drugs within one week that might affect the cardiovascular and neurological status

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | One month after the intervention
  Three ECG electrodes will beapplied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device (Mindray PM-8000 Express Patient Monitor, Bio-Medical Electricity, Hamburg, Germany). The ECG signals will be transferred to the PowerLab 16/30 (ADInstruments Pty Ltd. NSW, Australia) for data acquisition and analysis of the HRV.

SECONDARY OUTCOMES:
Heart rate | One month after the study
  Three ECG electrodes will be applied over left and right clavicles and left upper quadrant of abdomen respectively and then connect to a digital patient monitor device (Mindray PM-8000 Express Patient Monitor, Bio-Medical Electricity, Hamburg, Germany). The heart rate (HR) will be measured.

OTHER OUTCOMES:
Mean Blood pressure | One month afterwards
  Systolic and diastolic blood pressures will be taken on the left arm by a digital blood pressure monitor (Mindray PM-8000 Express Patient Monitor, Bio-Medical Electricity, Hamburg, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Tai Wai David Yu, MSc, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong, China